CLINICAL TRIAL: NCT00493948
Title: Evaluation of a Portable Device for Assessing Sleep Disordered Breathing in Congestive Heart Failure
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Rachel Coxon, ResMed
Other Study IDs: X06- 0237
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Heart Failure, Congestive; Sleep Apnea Syndromes
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ApneaLink — A two channel sleep screening device for the assessment of Sleep Disordered Breathing.

SUMMARY:
The purpose of this study is to evaluate an approved, portable device for assessing Sleep Disordered Breathing in Congestive Heart Failure.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe heart failure (as determined via Echocardiogram or treating physician)

Exclusion Criteria:

* Clinically significant asthma requiring therapy
* Significant (parenchymal) lung disease
* Severe pulmonary hypertension
* Hypercapnia (PCO2 > 60mmHg)
* Cardiogenic Shock
* Severe chronic renal failure
* Narcotic abuse/intravenous drug use (including heart failure due to alcohol abuse or chemotherapy, HIV+ and Hepatitis C)
* Methicillin- resistant Staphylococcus aureus infection
* Tracheotomy
* Enrolled in any concurrent study that may confound the results of this study
* Nocturnal positive airway pressure or oxygen
* Inability or refusal to sign patient consent form
* Inability or refusal to adhere to protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population under investigation are those people with moderate to severe heart failure who are currently admitted to the Coronary Care Unit of a major Sydney hospital.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2007-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Apnea- Hypopnea Index | Overnight

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Coxon, BE/MBiomedE, Study Director — ResMed/The University of New South Wales; Klaus Schindhelm, PhD, Study Director — ResMed/The University of New South Wales; Jodie Lattimore, PhD, Study Director — Royal Prince Alfred Hospital, Sydney, Australia; Ian Wilcox, PhD, Principal Investigator — Royal Prince Alfred Hospital/The University of Sydney
Locations (1):
- Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia